CLINICAL TRIAL: NCT02897128
Title: Transcutaneous Oxygen as a Predictor of Wound Healing Complications in Preoperatively Radiated Soft Tissue Sarcoma
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: University of Iowa (Other); University of Florida (Other); University of Oklahoma (Other); Orthopedic Research and Education Foundation (Other); Musculoskeletal Tumor Society (Unknown)
Responsible Party: Principal Investigator, Lukas Nystrom, MD, Associate Professor, Department of Orthopaedic Surgery, The Cleveland Clinic
Other Study IDs: 207638
Record Dates: First submitted 2016-09-07; First posted 2016-09-13 (Estimated); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Sarcoma, Soft Tissue
Keywords: Sarcoma; Radiation; Wound healing
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Observational Only - Transcutaneous Oxygen Measurement — The transcutaneous oxygen at your surgical site will be measured at three time points prior to your surgery.

SUMMARY:
Wound complications after sarcoma resection are frequent and potentially devastating problem. The burden of surgical wound complications in the lower extremity after preoperative external beam radiation therapy (EBRT) for soft tissue sarcoma is estimated at 43%. A noninvasive method of predicting complications would be extremely beneficial. The aim of this study is to evaluate the relationship between preoperative skin oxygenation and wound outcomes in a multi-center prospective analysis. This information could lead to a change in practice regarding surgical timing and adjunctive interventions to improve wound healing outcomes.

DETAILED DESCRIPTION:
It is estimated that there are 11,400 new cases of soft tissue sarcoma diagnosed in the United States annually. Most high-grade sarcomas, and other selected low or intermediate grade sarcomas, are treated with a limb salvage surgical resection in conjunction with external beam radiation to optimize local control. The current preference of most practicing orthopaedic/surgical oncologists and radiation oncologists is to implement the radiation treatments prior to surgery to diminish the total radiation dose and field size, thereby optimizing long-term functional results of the salvaged limb. While there are clear advantages of preoperative radiation, there are well-demonstrated negative consequences with regard to healing of the surgical wound. Currently there are no reliable clinical criteria to aid physicians in determining an individual patient's risk of developing a postoperative wound complication. This fact, combined with the rarity of the sarcoma diagnosis, has prevented improvement in wound outcomes in sarcoma patients.

This project is designed to close this critical gap in knowledge. The investigators propose utilizing a preoperative measurement of transcutaneous oxygen (Tc02) at the proposed incision to classify patients into high- and low-risk categories for development of wound complications after resection. Measurement of preoperative TcO2 represents a novel application of a simple, noninvasive method by which to assess skin oxygenation. Given the results of an already completed pilot investigation (Nystrom 2016), the investigators believe that this important clinical problem is well suited for a prospective, multi-disciplinary, multi-institutional investigation.

A successful project would result in an enhanced ability to identify wounds at risk prior to surgery and allow for additional investigation into perioperative interventions (delay of surgery until recovery of oxygenation, increasing suture duration, judicious use of muscle flaps and skin grafts, postoperative hyperbaric oxygen, or treatment with incisional wound vacuum-assisted closure) that may mitigate this significant adverse outcome.

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* biopsy proven soft tissue sarcoma of the lower extremity (pelvic area and below)
* plan for preoperative radiation and limb sparing resection

Exclusion Criteria:

* upper extremity sarcoma
* recurrent soft tissue sarcoma
* prior surgery in the area of the sarcoma
* prior radiation in the area of the sarcoma
* need for immediate skin graft or flap for coverage
* pregnant patients
* patients unwilling to have surgery or radiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with soft tissue sarcoma of the lower extremity with plan for treatment by preoperative radiation followed by limb sparing surgical resection.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2016-07; Primary Completion 2020-09-30 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Wound healing | 120 days
  Your wound will be assessed clinically for evidence of healing or any wound complication (ie. infection, dehiscence, seroma).

CONTACTS AND LOCATIONS:
Overall Officials: Lukas M Nystrom, MD, Principal Investigator — The Cleveland Clinic
Locations (4):
- United States (4):
  - University of Florida, Gainesville, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] O'Sullivan B, Davis AM, Turcotte R, Bell R, Catton C, Chabot P, Wunder J, Kandel R, Goddard K, Sadura A, Pater J, Zee B. Preoperative versus postoperative radiotherapy in soft-tissue sarcoma of the limbs: a randomised trial. Lancet. 2002 Jun 29;359(9325):2235-41. doi: 10.1016/S0140-6736(02)09292-9. PMID 12103287
- [Result] Nystrom LM, Miller BJ. Transcutaneous Oximetry May Predict Wound Healing Complications In Preoperatively Radiated Soft Tissue Sarcoma. Iowa Orthop J. 2016;36:117-22. PMID 27528847